CLINICAL TRIAL: NCT00960024
Title: Supported Employment for People With Severe Mental Illness in a Swedish Context- A Randomised Controlled Trial
Brief Title: Supported Employment in a Swedish Context
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Vardalinstitutet The Swedish Institute for Health Sciences (Other)
Responsible Party: Ulrika Bejerholm, the Vardal Institute, Medical Faculty, Lund University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: ulrika
Record Dates: First submitted 2009-08-14; First posted 2009-08-17 (Estimated); Last update posted 2009-08-17 (Estimated); Status verified 2009-08

CONDITIONS: Psychosis
Keywords: Vocational rehabilitation; Severe mental illness; Psychosis; Mental Health
MeSH Terms: conditions — Psychotic Disorders; Mental Disorders; Psychological Well-Being

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Individual Placement and Support-vocational rehabilitation (Experimental)
  Interventions: Behavioral: Individual Placement and Support-vocational rehabilitation
- Vocational rehabilitation available at study site (Active Comparator)
  Interventions: Behavioral: Vocational rehabilitation available

INTERVENTIONS:
Behavioral: Individual Placement and Support-vocational rehabilitation — Individual contact with an employment specialist, who works according to 7 core principles according to SE/IPS. 1) competitive employment as primary goal, 2) rapid job search, 3) eligibility based on client choice, 4) job search based on to client preferences, 5) integration with the mental health care team, 6) availability of time unlimited support at work 7) benefits counseling.
  Arms: Individual Placement and Support-vocational rehabilitation
Behavioral: Vocational rehabilitation available — The participants are offered vocational rehabilitation available at site
  Arms: Vocational rehabilitation available at study site

SUMMARY:
This project aims at generating evidence of a work-rehabilitation strategy that benefits the people with severe mental illness (SMI) who want to work, increase their sense of well-being and integration in society, decrease their financial dependence and experiences of stigma and discrimination. The project is likely to help form the basis of how to implement the evidence based supported employment (SE)-model, Individual Placement and Support model (IPS), in a Swedish work-rehabilitation context. In the long run, evidence of SE in a Swedish context could help to decrease the period of sick-leave and increase fulfilling and productive lifestyles among people with severe mental illness. In all, the effectiveness of SE can improve the quality of life for the target group, the quality in mental health care rehabilitation and decrease the costs of treatment and care.

DETAILED DESCRIPTION:
Evidence-based mental health treatment and scientific support has gained increased attention in Sweden. The Swedish National Board of Health and Welfare emphasizes the importance of Supported Employment. Especially since there are no study in Sweden that has an RCT-design, and that fully take on the responsibility of implementing a SE- intervention in concordance with the evidence based version of SE in mental health care, the Individual Placement and Support model, IPS. Internationally, SE according to IPS is an evidence-based approach to help people with SMI find and keep employment. RCT and quasi-experimental studies showed that IPS (Place-Then-Train), is more effective than the traditional stepwise vocational rehabilitation model(Train-Then-Place. However, there is no research evidence if the SE/IPS will function in relation to a Swedish benefit and health system and work-rehabilitation context. This intervention project will therefore not only study the effects of vocational and health-related outcomes and experiences, but also study the implementation of SE/IPS, its feasibility and level of fidelity in a Swedish context.

ELIGIBILITY:
Inclusion Criteria:

* People with Severe mental illness, which mostly means having a diagnosis of psychosis
* Communicate in Swedish
* Express interest in working in the near future
* Have professional care or support from psychiatric clinic
* Attend to a SE-introductory meeting

Exclusion Criteria:

* Additional organic or physical disability to having psychosis

Ages: 20 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Actual)
Dates: Start 2008-04; Primary Completion 2011-02 (Estimated); Study Completion 2015-12 (Estimated)

PRIMARY OUTCOMES:
To determine the effectiveness of SE/IPS in terms of vocational outcomes, such as employment rate, monthly income, job-tenure and working hours compared to stepwise rehabilitation available, for people with SMI in a Swedish context | 6 months, 18 months, and 24 months (6 months after end of intervention)

SECONDARY OUTCOMES:
To determine the effectiveness of a SE in terms health-related and functional outcomes, such as symptoms, perceived discrimination, empowerment, work-readiness, self-image, level of social and community participation, and quality of life | 6 months, 18 months, and 24 months (6 months after end of intervention)

CONTACTS AND LOCATIONS:
Overall Officials: Staffan Johansson, Assoc Prof, Study Director — Vardalinstitutet The Swedish Institute for Health Sciences
Locations (1):
- The Vardal Institute, Medical Faculty, Lund University, Lund, Sweden

REFERENCES:
- [Derived] Bejerholm U, Areberg C, Hofgren C, Sandlund M, Rinaldi M. Individual placement and support in Sweden - a randomized controlled trial. Nord J Psychiatry. 2015 Jan;69(1):57-66. doi: 10.3109/08039488.2014.929739. Epub 2014 Jul 1. PMID 24983382
- [Derived] Hasson H. Systematic evaluation of implementation fidelity of complex interventions in health and social care. Implement Sci. 2010 Sep 3;5:67. doi: 10.1186/1748-5908-5-67. PMID 20815872